CLINICAL TRIAL: NCT06300099
Title: Dexamethasone Versus Dexmedetomidine as Adjuncts to Serratus Anterior Plane Block for Postoperative Analgesia After Modified Radical Mastectomy A Randomized Clinical Study
Brief Title: Dexamethasone Versus Dexmedetomidine as Adjuncts to Serratus Anterior Plane Block
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Warda Demerdash Khalifa Ali, Principal investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AZAST/Research/52/20-Jan-2024
Record Dates: First submitted 2024-03-02; First posted 2024-03-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Dexamethasone; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Active Comparator): Dexamethasone injection
  Interventions: Drug: Dexamethasone
- Dexmedetomidine (Active Comparator): Dexmedetomidine injection.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone as adjunct to serratus anterior plane block.
  Arms: Dexamethasone
Drug: Dexmedetomidine — Dexmedetomidine as adjunct to serratus anterior plane block.
  Arms: Dexmedetomidine

SUMMARY:
Modified radical mastectomy is the most commonly performed surgical approach for breast cancer. The procedure enables surgeons to remove the main tumor mass, adjacent glandular tissue and regional lymph nodes. Moreover, it provides a cosmetic outcome that clearly surpasses the standard radical mastectomy and allows subsequent breast reconstruction with favorable results.

The present randomized study aims to compare the postoperative analgesic effects of dexamethasone and dexmedetomidine as adjuncts to serratus anterior plane block in women undergoing modified radical mastectomy.

DETAILED DESCRIPTION:
Modified radical mastectomy is the most commonly performed surgical approach for breast cancer. The procedure enables surgeons to remove the main tumor mass, adjacent glandular tissue and regional lymph nodes. Moreover, it provides a cosmetic outcome that clearly surpasses the standard radical mastectomy and allows subsequent breast reconstruction with favorable results.

Serratus anterior plane block (SAPB) with ultrasound guidance is a fascial plane block that proved to be feasible, safe and effective tool for reduction of postoperative pain after thoracic and breast surgeries. In multiple instances, SAPB is used with additional adjuncts e.g. dexamethasone or dexmedetomidine to improve analgesic potency and duration.

ELIGIBILITY:
Inclusion Criteria:

Consecutive American Society of Anesthesiologists (ASA) class I-II female patients with breast cancer indicated for modified radical mastectomy

Exclusion Criteria:

Allergy to the study medications . Patients will also be excluded if they have history of chronic pain conditions, opioid dependence or if they received prolonged analgesic therapy prior to surgery.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 126 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
postoperative visual assessment scale for pain. | 72 hours postoperative
  Subjective pain assessment scale

IPD SHARING:
Plan to Share IPD: No